CLINICAL TRIAL: NCT04650490
Title: A Randomized, Phase II Trial of SRS Timing With Immune Checkpoint Inhibition in Patients With Untreated Brain Metastases From Non-small Cell Lung Cancer
Brief Title: SRS Timing With Immune Checkpoint Inhibition in Patients With Untreated Brain Metastases From Non-small Cell Lung Cancer
Acronym: STICk-IM-NSCLC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: failure to enroll
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00106340
Record Dates: First submitted 2020-11-17; First posted 2020-12-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Brain Metastases; Non Small Cell Lung Cancer
Keywords: immunotherapy; Stereotactic radiosurgery
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate SRS followed by IO (Experimental): Participants will receive SRS followed by physician's choice of standard of care immunotherapy, given at the FDA-approved dose within 14 days of SRS.
  Interventions: Radiation: Stereotactic Radiosurgery; Drug: Immunotherapy
- Immediate IO followed by SRS (Experimental): Participants will receive physician's choice of immunotherapy, given at the FDA-approved dose followed by SRS, if deemed appropriate, at the time of intracranial progression.
  Interventions: Radiation: Stereotactic Radiosurgery; Drug: Immunotherapy

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — Timing of stereotactic radiosurgery relative to immunotherapy
Drug: Immunotherapy — Physician's choice of immunotherapy per standard of care

SUMMARY:
This trial is a randomized, 2-arm, phase II study to determine the effect, if any, of the timing of stereotactic radiosurgery (SRS) relative to immune checkpoint inhibitor (IO) therapy in patients with non-small cell lung cancer (NSCLC) that has spread (metastasized) to the brain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have 1 to 15 newly diagnosed brain metastases, ≤5 cm in the largest dimension, with at least one metastasis measuring ≥0.3 cm.
2. Primary tumor histology must be one confirmed as one of the following:

   1. Squamous NSCLC
   2. Adenocarcinoma NSCLC
   3. Not otherwise specified NSCLC
3. Patient must have an MRI of the brain within 4 weeks (28 days) of signing the study consent.
4. Patient must be planned for immunotherapy treatment as their next systemic therapy, including monotherapy or in combination with chemotherapy.
5. Patients previously treated with a tyrosine kinase inhibitor (TKI) may be eligible, if a second line (or later) immunotherapy regimen is planned.
6. Patients must be asymptomatic or minimally symptomatic, requiring the equivalent of ≤2 mg dexamethasone/day for at least 7 days prior to enrollment.
7. Female and male subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in the Duke Contraception Policy.
8. Age ≥18 years of age at the time of entry into the study.
9. Karnofsky Performance Score (KPS) ≥70.

Exclusion Criteria:

1. Patients on the equivalent of >2 mg of dexamethasone (or prednisone/steroid equivalent) daily ≤ 7 days before receiving study treatment.
2. Patients who have previously received whole brain radiation therapy (WBRT).
3. Patients must not have ever received immunotherapy in the stage IV setting. Prior immune therapy as part of treatment for stage I-III disease is allowed after an interval of >6 months has passed from the completion of that therapy.
4. Patients with leptomeningeal carcinomatosis. However, patients with discrete dural-based lesions may be eligible at the discretion of the treating radiation oncologist.
5. Females who are pregnant or breastfeeding.
6. Patients with an impending, life-threatening cerebral hemorrhage or herniation, based on the assessment from a brain MRI of the study neurosurgeons or their designee.
7. Patients with severe, active co-morbidity, defined as follows:

   1. Patients with an active infection requiring intravenous treatment or having an unexplained febrile illness (Tmax > 99.5°F/37.5°C)
   2. Patients with known immunosuppressive disease or known uncontrolled human immunodeficiency virus infection
   3. Patients with unstable or severe intercurrent medical conditions such as severe heart disease (New York Heart Association Class 3 or 4)
8. Patients who have not recovered from the toxic effects of prior chemo- and/or radiation therapy. Guidelines for this recovery period are dependent upon the specific therapeutic agent being used.
9. Patients with prior, unrelated malignancy requiring current active treatment in the last 3 years with the exception of cervical carcinoma in situ, prostate cancer at stage I-III and adequately treated basal cell or squamous cell carcinoma of the skin
10. Patients with a known history of hypersensitivity to the physician's choice of immune checkpoint inhibitor, or any components of the inhibitor.
11. Patients who have any contraindications to immunotherapy.
12. Patients with active autoimmune disease requiring systemic immunomodulatory treatment, including steroid of >10 mg prednisone daily or equivalent, within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Intracranial progression free-survival | from randomization through study completion, an average of 3 years
  Defined as defined as time to intracranial progression from randomization measured by by RANO-BM criteria for radiographic progression on contrast-enhanced brain MRI

SECONDARY OUTCOMES:
Assess quality of life in each arm by the Functional Assessment of Cancer Therapy - Brain questionnaire | 1 year
  as measured on a 5 point Likert-type scale from 0 (not at all) through 4 (very much) where the higher score reflects better quality of life
Assess neurocognitive outcome in each arm by the Hopkins Verbal Learning Test - Revised | 1 year
  as measured by recall scores with higher values indicating better outcomes
Assess neurocognitive outcome in each arm by the Trail Making Test Parts A and B | 1 year
  scored as average or deficient based on time to complete the activity
Assess neurocognitive outcome in each arm by the Controlled Oral Word Association test | 1 year
  scored as the number of words completed in one minute, with higher score indicating better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Scott Floyd, MD PhD, Principal Investigator — Duke Health; Jeffrey Clarke, MD, Principal Investigator — Duke Health
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No